CLINICAL TRIAL: NCT04889703
Title: A Pilot Study Testing the Effects of Chemical Peels in Patients With Rosacea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Plan to move forward with this study has been dropped
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heather Woodworth Goff, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0804
Record Dates: First submitted 2021-04-27; First posted 2021-05-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15% Trichloroacetic acid (TCA) chemical peel (Experimental): 15% trichloroacetic acid will be applied topically on the skin of the entire face in two separate clinic visits that are 4 weeks apart
  Interventions: Drug: 15% Trichloroacetic acid peel
- 30% Salicylic acid chemical peel (Experimental): 30% salicylic acid will be applied topically on the skin of the entire face in two separate clinic visits that are 4 weeks apart
  Interventions: Drug: 30% Salicylic acid peel

INTERVENTIONS:
Drug: 15% Trichloroacetic acid peel — Trichloroacetic acid peel (15%) will be applied topically to the face for 2 treatments at 4 week intervals.
  Arms: 15% Trichloroacetic acid (TCA) chemical peel
Drug: 30% Salicylic acid peel — Salicylic acid peel (30%) will be applied topically to the face for 2 treatments at 4 week intervals.
  Arms: 30% Salicylic acid chemical peel

SUMMARY:
The study is a prospective, randomized, one-site therapeutic trial of 15% trichloroacetic acid (TCA) and 30% salicylic acid peels for rosacea. Two peels will be applied topically 4 weeks apart, and the study will end in 12 weeks. Endpoints include adverse affects within the first 8 weeks and responses, which will be measured by Investigator Global Assessment (IGA), a Rosacea Clinical Scorecard, and number of papular plus pustular lesions assessed every 4 weeks up to 12 weeks with high resolution photographs.

Treatment Dosage and administration

Study Drugs:

1. Trichloroacetic acid peel (15%) will be applied topically to the face for 2 treatments at 4 week intervals.
2. Salicylic acid peel (30%) will be applied topically to the face for 2 treatments at 4 week intervals.

Duration of treatment: two single applications 4 weeks apart.

Endpoint: 12 weeks after first chemical peel treatment

Outcome measures:

* independent objective reviewer scoring of matched photographs before and after treatment
* number of papular and pustular lesions before and after treatment
* rosacea-specific patient quality of life survey responses before and after treatment

  * Adverse effects such as peeling, redness, scaling, crusting, blister formation, and hyperpigmentation will be assessed clinical

DETAILED DESCRIPTION:
Patients with a diagnosis of rosacea will be included. Peels will be performed at no cost to participants; funding will be supplied by the UT Southwestern Dermatology department. A total of 20 patients will be consented. At the initial visit, patients will fill out a form with demographic information as well as a RosaQOL survey about how their rosacea has affected their quality of life. High-quality photographs of each patient's baseline rosacea will be taken. The treatment arms of 15% TCA peel and 30% salicylic acid peel will be randomly assigned to patients, and the topical treatment will be applied to the entire face. The duration of involvement of each subject from the time of initial consent to final clinical evaluation will be 12 weeks. There will be a total of 4 clinical visits lasting approximately 30 minutes per visit. Each patient will undergo two chemical peel treatments, with a 4-week interval between treatments. The first treatment will occur at 0 weeks (first visit). Each patient will follow up at 4 weeks (second visit) for his or her second chemical peel treatment. After two treatments, the patient will then follow up at 8 weeks (third visit) and 12 weeks (fourth visit) for evaluation of response to treatment.

For the chemical peel treatment, each patient's face will be prepared by cleansing with a deep cleanser, followed by removal of sebum utilizing either alcohol or acetone as a degreasing agent, and allowing the skin to dry. These steps help optimize penetration of the peeling agent. The peeling agent will then be applied uniformly to the face with a 2X2 gauze pad with the patient in supine position until adequate erythematous response is observed. If needed, the acidic peeling agent may be neutralized with water. Patients will be instructed to apply Vaseline and sunscreen to the face daily post-treatment to keep the skin moisturized and protected from UV radiation until exfoliation is complete, typically within 7-10 days post-peel.

The outcome measures will include patient quality of life survey responses, independent objective reviewer scoring of matched photographs, and comparisons of the number of papular and pustular lesions before and after treatment. At each visit, the total number of papular and pustular lesions will be recorded. High resolution photographs of both the left and right sides of the face will be taken at the first visit to serve as each patient's baseline rosacea. Patients will also be asked to complete the RosaQOL survey at the first clinical visit. Additional photographs will be taken at all four visits using identical lighting, positioning, and settings for all patients. Two independent investigators will score matched photographs of the baseline and treated rosacea at time points 0 weeks, 8 weeks, and 12 weeks using a scale from 0 to 6. 0 indicates no papules, pustules, residual erythema, or telangiectasia; 1 indicates rare papules and/or pustules, residual to mild erythema, and mild to moderate telangiectasia; 2 indicates few papules and/or pustules, mild erythema, and mild to moderate telangiectasia; 3 indicates a distinct number of papules and/or pustules, mild to moderate erythema, and mild to moderate telangiectasia; 4 indicates a pronounced number of papules and/or pustules, moderate erythema, and mild to moderate telangiectasia; 5 indicates many papules and/or pustules occasionally with large inflamed lesions, moderate erythema, and moderate telangiectasia; and 6 indicates numerous papules and/or pustules occasionally with confluent areas of inflamed lesions, moderate or severe erythema, and moderate or severe telangiectasia16. Independent observer scores will be graded using the same method and same scale for all patients.

At the 12-week follow up visit, patients will be asked to repeat the RosaQOL survey. Photographs will be taken, and a final documentation of gross number of papular and pustular lesions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rosacea, with both papular/pustular lesions and facial erythema

Exclusion Criteria:

* patients with active skin infection involving the face
* patients with severe nodular or phymatous rosacea with ocular involvement
* patients with other dermatoses that may interfere with the evaluation of rosacea
* patients who are pregnant or breastfeeding
* use of isotretinoin within the last year
* history of hypersensitivity to chemical peeling
* patients who easily scar or have dyspigmentation tendencies
* patients who continue to experience excessive sun exposure
* patients planning to change or initiate other treatments for their rosacea during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Independent objective reviewer scoring of matched photographs | Done at 0 weeks of study
  Two independent investigators will score matched photographs of the baseline rosacea at time point 0 weeks using a scale from 0 to 6. 0 indicates no papules, pustules, residual erythema, or telangiectasia; 1 indicates rare papules and/or pustules, residual to mild erythema, and mild to moderate telangiectasia; 2 indicates few papules and/or pustules, mild erythema, and mild to moderate telangiectasia; 3 indicates a distinct number of papules and/or pustules, mild to moderate erythema, and mild to moderate telangiectasia; 4 indicates a pronounced number of papules and/or pustules, moderate erythema, and mild to moderate telangiectasia; 5 indicates many papules and/or pustules occasionally with large inflamed lesions, moderate erythema, and moderate telangiectasia; and 6 indicates numerous papules and/or pustules occasionally with confluent areas of inflamed lesions, moderate or severe erythema, and moderate or severe telangiectasia.
Independent objective reviewer scoring of matched photographs | Done at 4 weeks of study
  Two independent investigators will score matched photographs of the baseline rosacea at time point 4 weeks using a scale from 0 to 6. 0 indicates no papules, pustules, residual erythema, or telangiectasia; 1 indicates rare papules and/or pustules, residual to mild erythema, and mild to moderate telangiectasia; 2 indicates few papules and/or pustules, mild erythema, and mild to moderate telangiectasia; 3 indicates a distinct number of papules and/or pustules, mild to moderate erythema, and mild to moderate telangiectasia; 4 indicates a pronounced number of papules and/or pustules, moderate erythema, and mild to moderate telangiectasia; 5 indicates many papules and/or pustules occasionally with large inflamed lesions, moderate erythema, and moderate telangiectasia; and 6 indicates numerous papules and/or pustules occasionally with confluent areas of inflamed lesions, moderate or severe erythema, and moderate or severe telangiectasia.
Independent objective reviewer scoring of matched photographs | Done at 8 weeks of study
  Two independent investigators will score matched photographs of the baseline rosacea at time point 8 weeks using a scale from 0 to 6. 0 indicates no papules, pustules, residual erythema, or telangiectasia; 1 indicates rare papules and/or pustules, residual to mild erythema, and mild to moderate telangiectasia; 2 indicates few papules and/or pustules, mild erythema, and mild to moderate telangiectasia; 3 indicates a distinct number of papules and/or pustules, mild to moderate erythema, and mild to moderate telangiectasia; 4 indicates a pronounced number of papules and/or pustules, moderate erythema, and mild to moderate telangiectasia; 5 indicates many papules and/or pustules occasionally with large inflamed lesions, moderate erythema, and moderate telangiectasia; and 6 indicates numerous papules and/or pustules occasionally with confluent areas of inflamed lesions, moderate or severe erythema, and moderate or severe telangiectasia.
Independent objective reviewer scoring of matched photographs | Done at 12 weeks of study
  Two independent investigators will score matched photographs of the baseline rosacea at time point 12 weeks using a scale from 0 to 6. 0 indicates no papules, pustules, residual erythema, or telangiectasia; 1 indicates rare papules and/or pustules, residual to mild erythema, and mild to moderate telangiectasia; 2 indicates few papules and/or pustules, mild erythema, and mild to moderate telangiectasia; 3 indicates a distinct number of papules and/or pustules, mild to moderate erythema, and mild to moderate telangiectasia; 4 indicates a pronounced number of papules and/or pustules, moderate erythema, and mild to moderate telangiectasia; 5 indicates many papules and/or pustules occasionally with large inflamed lesions, moderate erythema, and moderate telangiectasia; and 6 indicates numerous papules and/or pustules occasionally with confluent areas of inflamed lesions, moderate or severe erythema, and moderate or severe telangiectasia.

SECONDARY OUTCOMES:
Total number of papular and pustular lesions | Done at 0 weeks of study
  The total number of papular and pustular lesions will be recorded by the researcher.
Total number of papular and pustular lesions | Done at 4 weeks of study
  The total number of papular and pustular lesions will be recorded by the researcher.
Total number of papular and pustular lesions | Done at 8 weeks of study
  The total number of papular and pustular lesions will be recorded by the researcher.
Total number of papular and pustular lesions | Done at 12 weeks of study
  The total number of papular and pustular lesions will be recorded by the researcher.
Rosacea Quality of Life (QOL) Survey Response | Completed by patient at 0 weeks of study
  Patients will be asked to complete a rosacea-specific quality of life survey before the initiation of treatment to measure thoughts about their baseline rosacea. Answers are based on a scale from 1-5 and are quantifiable.
Rosacea Quality of Life (QOL) Survey Response | Completed by patient at 12 weeks of study
  Patients will be asked to complete a rosacea-specific quality of life survey after completion of treatment to measure thoughts about their rosacea. Answers are based on a scale from 1-5 and are quantifiable.

IPD SHARING:
Plan to Share IPD: No